CLINICAL TRIAL: NCT01591213
Title: St. Jude Cancer Education for Children Program: The Feasibility of Teacher Delivery (Pilot Study)
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XPD12-040 SJCECP2
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Cancer education; Prevention education; Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Fourth grade students enrolled in Memphis-area schools.

SUMMARY:
-The St. Jude Cancer Education for Children Program was created in 2006 as part of the outreach mandate of the Comprehensive Cancer Center at St. Jude Children's Research Hospital. The curriculum is designed to teach schoolchildren about cancer and dispel common misconceptions, inform students about healthy lifestyle choices that can translate to reduced cancer risk in adulthood, and to inspire an interest in science and scientific careers. In the 2010-2011 school year, researchers examined the impact of the program in regard to knowledge.

It has always been clear that St. Jude personnel are limited to visiting a small number of schools in person each year so in 2011, a teacher's kit to the education program was created. The kit includes all the lesson plans needed to complete the program without the presence of St. Jude staff members. As a result, researchers at St. Jude Children's Research Hospital want to test the feasibility of the intervention by schoolteachers, and how this mechanism of delivery will affect student knowledge, attitudes, and health behaviors associated with cancer and healthy living.

DETAILED DESCRIPTION:
Teachers who agree to participate will use the teacher's kit developed by the St. Jude International Outreach Program to deliver the St. Jude Cancer Education for Children curriculum to 4th grade students over the course of 1 week. Pre and post survey data will be collected from students to measure knowledge, beliefs, attitudes, perceptions of vulnerability, intentions, and behaviors associated with cancer and healthy living. Rates of compliance and feedback about the curriculum will be collected from teachers via curriculum checklist, survey, and interviews.

Primary Objective:

* To determine if it is feasible for classroom teachers to implement the St. Jude Cancer Education for Children Program.

Secondary/Exploratory Objectives:

* To determine factors that may contribute to the program's feasibility such as school and teacher characteristics.
* To measure the impact of the intervention on student knowledge, beliefs, attitudes, perceptions of vulnerability, intentions, and self-reported health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Located in the United States or United States territories
* District & school provide permission
* 3rd, 4th, or 5th grade student with cognitive capacity to complete questionnaires (as determined by the teacher)
* Assents to study participation

Exclusion Criteria:

* Located outside of the United States or United States territories
* Student does not assent to participation
* Student without cognitive capacity to complete questionnaires (as determined by the teacher)
* Parent or guardian refuses consent

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fourth grade students enrolled in Memphis-area schools.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Rate of compliance | 1 week (at end of three teaching modules)
  Delivery of the educational curriculum by classroom teachers will be demonstrated to be a feasible method of delivering the St. Jude Cancer Education for Children Program. The program will be determined to be feasible if 80% of the schools that agree to participate complete the delivery of the program. A complete delivery will be defined as all grade consenting teachers delivering 2/3 of the educational content in each of the three modules.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Ayers, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols